CLINICAL TRIAL: NCT05434468
Title: Comparative Effects of Sustained Neutral Apophyseal Glides Half Rotation Technique and Gong's Mobilizations in Cervicogenic Headache
Brief Title: Sustained Neutral Apophyseal Glides Half Rotation Technique and Gong's Mobilizations in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0133
Record Dates: First submitted 2022-04-15; First posted 2022-06-28 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Cervicogenic Headache
Keywords: cervicogenic headache ,Gong's mobilization ,
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained neutral apophyseal glides group (Experimental): Sustained neutral apophyseal glides will apply on this group.
  Interventions: Other: Sustained neutral apophyseal glides
- Gong mobilization (Experimental): mobilization technique
  Interventions: Other: Sustained neutral apophyseal glides

INTERVENTIONS:
Other: Sustained neutral apophyseal glides — gong mobilization
  Other Names: gong mobilization

SUMMARY:
Cervicogenic headache is a very incessant issue that is often faced by general population.Cervicogenic headache is a significant issue in patients with upper cervical dysfunction. However, its physical therapy management is a subject of debate.As the Comparative effects of SNAGs half rotation technique and Gong's mobilizations has never been investigated in patients with cervicogenic headache and neck pain , the aim of this study is to investigate the effects of these treatments on two study groups(Group A&B) respectively. This study will be a randomized clinical trial and will be conducted in D.H.Q Sahiwal . The study will be completed within the time duration of six months .Non- probability convenience sampling technique will be used to collect the data. The sample size of 30 patients will be taken in this study , aged 25-45 years, will allocate to two groups, Group A (Sustained neutral apophyseal glide half rotation technique) Group B (Gong's mobilization).cervical Sustained neutral apophyseal glide half rotation technique (SNAG) half rotation technique will be performed with the patient sitting on a chair in the erect posture. The thumb placement of therapist will be over the transverse process of C1. Then, glide will be applied ventrally with active rotation of the restricted site 10 times holding for 10 seconds with overpressure at end of the rotation with 30 second rest in between each repetition and 3 session/week for 6 weeks.Group B will be treated three times in a week for 4 weeks.Group B will get Gong's mobilization for 15-20 mins.Participants will be treated 3 times per week for 6 weeks. Pre and Post treatment readings will be taken in 1st session and 6th week respectively. Assessment will done via flexion rotation test (FRT),6-item Headache Impact scale and neck disability index. Neck Disability Index will use to examine neck pain intensity and cervicogenic headache symptoms.

DETAILED DESCRIPTION:
Cervicogenic headache is a very incessant issue that is often faced by general population.Cervicogenic headache is a significant issue in patients with upper cervical dysfunction. However, its physical therapy management is a subject of debate.As the Comparative effects of SNAGs half rotation technique and Gong's mobilizations has never been investigated in patients with cervicogenic headache and neck pain , the aim of this study is to investigate the effects of these treatments on two study groups(Group A&B) respectively. This study will be a randomized clinical trial and will be conducted in D.H.Q Sahiwal . The study will be completed within the time duration of six months .Non- probability convenience sampling technique will be used to collect the data. The sample size of 30 patients will be taken in this study , aged 25-45 years, will allocate to two groups, Group A (Sustained neutral apophyseal glide half rotation technique) Group B (Gong's mobilization).cervical Sustained neutral apophyseal glide half rotation technique (SNAG) half rotation technique will be performed with the patient sitting on a chair in the erect posture. The thumb placement of therapist will be over the transverse process of C1. Then, glide will be applied ventrally with active rotation of the restricted site 10 times holding for 10 seconds with overpressure at end of the rotation with 30 second rest in between each repetition and 3 session/week for 6 weeks.Group B will be treated three times in a week for 4 weeks.Group B will get Gong's mobilization for 15-20 mins.Participants will be treated 3 times per week for 6 weeks. Pre and Post treatment readings will be taken in 1st session and 6th week respectively. Assessment will done via flexion rotation test (FRT),6-item Headache Impact scale and neck disability index. Neck Disability Index will use to examine neck pain intensity and cervicogenic headache symptoms. The 6-item Headache Impact Test scale will use to examine headache severity and its adverse effects on social life and functions. Flexion-Rotation Test will use to assess rotation range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Headache with neck stiffness and pain.
* Headache for the past 3 months at least once per week
* Aged 25-45 years
* Chronic neck pain for more than 3 months
* baseline NDI score of atleast

Exclusion Criteria:

* Physiotherapy or chiropractic treatment in the past 3 months
* Headache with autonomic involvement, dizziness, or visual disturbance
* Congenital conditions of the cervical spine
* Contraindication to manipulative therapy
* Involvement in litigation or compensation
* Inability to tolerate the flexion-rotation test

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
neck disablity index | 6 months
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. ... A higher NDI score means the greater a patient's perceived disability due to neck pain. The minimally clinically important change by patients has been found to be 5 or 10%.
flexion rotation test | 6 months
  The passive flexion-rotation test (FRT-P) is performed with the patient supine. An examiner passively positions the patient's neck into full flexion to pre-tension the structures of the middle and lower cervical spine, then the patient's head is passively rotated each direction while the flexed position is maintained.
HIT questionnaire | 6 months
  The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the
goniometer | 6 months
  for measuring range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, PhD, Study Chair — Riphah International University
Locations (1):
- Railway Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ylinen J, Nikander R, Nykanen M, Kautiainen H, Hakkinen A. Effect of neck exercises on cervicogenic headache: a randomized controlled trial. J Rehabil Med. 2010 Apr;42(4):344-9. doi: 10.2340/16501977-0527. PMID 20461336
- [Background] Mohamed AA, Shendy WS, Semary M, Mourad HS, Battecha KH, Soliman ES, Sayed SHE, Mohamed GI. Combined use of cervical headache snag and cervical snag half rotation techniques in the treatment of cervicogenic headache. J Phys Ther Sci. 2019 Apr;31(4):376-381. doi: 10.1589/jpts.31.376. Epub 2019 Apr 1. PMID 31037013